CLINICAL TRIAL: NCT00334217
Title: Cognitive Remediation in the Initial Phase of Substance Abuse Treatment: Feasibility and Efficacy
Brief Title: Cognitive Remediation in Early Substance Abuse Treatment
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The intervention could not be successfully carried out in the SADP setting because of issues independent of the cognitive training intervention.
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Bell, Morris - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: O3108R
Record Dates: First submitted 2006-06-02; First posted 2006-06-06 (Estimated); Last update posted 2009-06-18 (Estimated); Status verified 2009-06

CONDITIONS: Substance-Related Disorders
Keywords: Psychology: cognitive aspects; Substance-Related Disorders; treatment efficacy
MeSH Terms: conditions — Substance-Related Disorders | interventions — Cognitive Remediation

ARMS (2):
- 1 (Experimental): PSS CogRehab exercises
  Interventions: Behavioral: Cognitive Remediation
- 2 (No Intervention): On-line computer games

INTERVENTIONS:
Behavioral: Cognitive Remediation — PSS Cogrehab
  Arms: 1

SUMMARY:
This study is for the purpose of determining whether cognitive remediation may improve cognition and treatment response in patients entering substance abuse day treatment

DETAILED DESCRIPTION:
Background: Patients entering substance abuse treatment display cognitive deficits that may reduce their ability to benefit from their treatment. While there is considerable variety in the severity and types of cognitive impairment found in newly recovering patients, problems with attention, memory and executive function are very common. Since treatment requires sustained attention, remembering what is learned, integrating that knowledge and applying it to recovery, impairment in underlying cognitive processes makes successful treatment less likely. Although cognitive functioning improves with sustained sobriety, it is during the early phase of recovery that most patients receive the most intensive treatment. Recent research has suggested that cognitive remediation exercises during this early phase may speed up the return of cognitive functioning and in so doing may have a direct effect on whether patients find the treatment useful and complete their treatment. By keeping patients in treatment longer, cognitive remediation may have an indirect effect on substance abuse outcomes.

Objectives: To pilot test the introduction of cognitive remediation at the Substance Abuse Day Treatment Program (SADP) at the Errara Community Care Center. Aims are 1) to assess the receptivity of patients to the intervention by determining rates of agreement to participate, 2) to determine the number of cognitive remediation sessions that patients are willing to engage in, 3) to assess a variety of cognitive remediation tasks for their acceptability, 4) to evaluate neuropsychological improvements using pre-post assessment, 5) to evaluate its effects on substance abuse treatment participation, and 6) to evaluate its effects on substance abuse outcomes at 6 months follow-up.

Design: Randomized clinical trial of cognitive remediation with an active control condition with observations at baseline, end of treatment and 6-months from intake

ELIGIBILITY:
Inclusion Criteria:

* Veterans participating in a substance abuse day treatment program at the Errara Community Center

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2005-08; Primary Completion 2007-08 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Cognitive improvement and adherence to substance abuse treatment | 6 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Morris D Bell, PhD, Principal Investigator — VA Connecticut Health Care System (West Haven)
Locations (1):
- VA Connecticut Health Care System (West Haven), West Haven, Connecticut, United States

REFERENCES:
- [Result] Horner MD, Harvey RT, Denier CA. Self-report and objective measures of cognitive deficit in patients entering substance abuse treatment. Psychiatry Res. 1999 May 31;86(2):155-61. doi: 10.1016/s0165-1781(99)00031-1. PMID 10397417
- [Result] Teichner G, Horner MD, Roitzsch JC, Herron J, Thevos A. Substance abuse treatment outcomes for cognitively impaired and intact outpatients. Addict Behav. 2002 Sep-Oct;27(5):751-63. doi: 10.1016/s0306-4603(01)00207-6. PMID 12201382
- [Result] Grohman K, Fals-Stewart W. The detection of cognitive impairment among substance-abusing patients: the accuracy of the neuropsychological assessment battery-screening module. Exp Clin Psychopharmacol. 2004 Aug;12(3):200-7. doi: 10.1037/1064-1297.12.3.200. PMID 15301637
- [Result] O'Malley S, Adamse M, Heaton RK, Gawin FH. Neuropsychological impairment in chronic cocaine abusers. Am J Drug Alcohol Abuse. 1992;18(2):131-44. doi: 10.3109/00952999208992826. PMID 1562011